CLINICAL TRIAL: NCT05752253
Title: Counseling Intervention in Hereditary Hemorrhagic Telangiectasia in the COVID Era.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mazza Marianna, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3136
Record Dates: First submitted 2023-02-26; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Hereditary Hemorragic Teleangectasia (Other): Patients with Hereditary Hemorragic Teleangectasia
  Interventions: Other: Counseling

INTERVENTIONS:
Other: Counseling — Counseling is a process which, through positive orientation and the enhancement of personal resources, is aimed at promoting the improvement of the quality of life in the other.

SUMMARY:
The goal of this interventional study is to determine the incidence of depression, anxiety, sleep disturbances and resilience in a sample of subjects affected by Hereditary Hemorrhagic Telangiectasia. The study is declined through the evaluation of some outcome parameters at the time of enrollment (T0), during the counseling intervention (T1 and T2) and at the end (T3) of the subjects who will have carried out an individual counseling intervention.

ELIGIBILITY:
Inclusion Criteria:

Recruited subjects have a diagnosis of Hereditary Hemorrhagic Telangiectasia and are 18 years of age or older.

Exclusion Criteria:

Previous or current intellectual disability and a diagnosis of psychiatric disorders in accordance with the Diagnostic and Statistical Manual of Mental Disorders, DSM-5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Administration of psychometric scales
Connor-Davidson Resilience Scale (CD-RISC) | 12 months
  Administration of psychometric scales
Pittsburgh Sleep Quality Index (PSQI); | 12 months
  Administration of psychometric scales

SECONDARY OUTCOMES:
Impact of counseling on clients affected by rare diseases | 12 months
  Administration of psychometric scales

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No